CLINICAL TRIAL: NCT02470728
Title: Pain Management Options for Opioid Tolerant Patients: a Randomized Controlled Trial
Brief Title: Optimal Management of Pain in Hospitalized Patients - Opioid Tolerant Populations.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary issues
Sponsor: Duke University (Other)
Collaborators: Massachusetts Institute of Technology (Other); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00076402
Record Dates: First submitted 2015-01-13; First posted 2015-06-12 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pain; Acute Pain; Postoperative Pain
Keywords: patient readmission; pain relief units; pain centers; multidisciplinary pain clinics; multidisciplinary pain centers; pain clinics; hospital readmission; emergencies; emergency medicine; critical care; emergency treatment; opioid; acute pain service
MeSH Terms: conditions — Pain; Acute Pain; Pain, Postoperative; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Those randomized into the control group will receive the current standard of care for pain management. This standard care pathway involves a pain management specialist consultation only at the request of the primary admitting team. The pain management consultation can occur at any time during the patient's inpatient stay and care by these specialists ends at discharge.
- Treatment Group (Experimental): Subjects randomized into the treatment (early intervention) group will receive the New Clinical Pathway: pain management care coordinated by pain-management specialists from inpatient admission through 60 days after discharge.
  Interventions: Other: New Clinical Pathway

INTERVENTIONS:
Other: New Clinical Pathway
  Arms: Treatment Group

SUMMARY:
Pain is a symptom that drives hospital admissions, and pain management is required by most patients during their hospital stay. Further, the use of medications such as opioids can lead to upward-spiraling doses, especially among chronic pain patients whose resource utilization rates are high. Many initiatives aim to reduce the costs of these "high-resource utilizing" patients. One exciting aspect of improving the management of pain is that this may help prevent patients from ever becoming high-cost in the first place. The purpose of this study is to examine the impacts of an early and sustained intervention pathway, in comparison to the current standard of care, for the treatment of pain in opioid tolerant patients. It is hypothesized that patients randomized to the intervention pathway, in comparison to the control, will lead to decreased costs of care, a reduction in opioid usage within 3 and 6 months, and decrease in hospital readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Known opioid tolerant (as determined per FDA criteria)
* Agree to sign the informed consent and HIPAA forms

Exclusion Criteria:

* Patients under the age of 18 years
* No known opioid tolerance
* Do not agree to sign the informed consent and HIPAA forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Returns to Acute Care | Discharge through 90 days post-discharge
  Hospital Readmissions and Emergency Department Utilizations

SECONDARY OUTCOMES:
Opioid Analgesic Use | Discharge through 90 days post-discharge
  Quantification of opioid analgesic use over time
Opioid Analgesic Use | Admission through 12 months post-discharge
  Quantification of opioid analgesic use over time
Opioid Tolerance Status | Admission through 12 months post-discharge
  Opioid tolerance as inferred from opioid prescription and usage per FDA exposure threshold definition for opioid tolerance.
Pain at Discharge | Measured upon day of discharge from index hospitalization; up to 18 months from the date of randomization
  Patient-reported pain at the time of discharge from index hospitalization
Hospital Length of Stay | Measured upon day of discharge from index hospitalization; up to 18 months from the date of randomization
  Duration of index inpatient hospitalization.
Latency to Hospital Readmission | Discharge through 12 months post-discharge
  Time between discharge from index hospitalization to readmission
Returns to Acute Care | Discharge through 12 months post-discharge
  Hospital Readmissions and Emergency Department Utilizations at an extended time horizon
Healthcare Expenditures | Admission through 12 months post-discharge
  Inpatient and outpatients costs
Use of Rescue Drugs | Admission through 12 months post-discharge
  Antagonist usages for the reversal of index drug effects (opioid and benzodiazepine)

CONTACTS AND LOCATIONS:
Overall Officials: Padma Gulur, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of California, Irvine Medical Center, Orange, California
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Raebel MA, Newcomer SR, Reifler LM, Boudreau D, Elliott TE, DeBar L, Ahmed A, Pawloski PA, Fisher D, Donahoo WT, Bayliss EA. Chronic use of opioid medications before and after bariatric surgery. JAMA. 2013 Oct 2;310(13):1369-76. doi: 10.1001/jama.2013.278344. PMID 24084922
- [Background] Brown EG, Burgess D, Li CS, Canter RJ, Bold RJ. Hospital readmissions: necessary evil or preventable target for quality improvement. Ann Surg. 2014 Oct;260(4):583-9; discussion 589-91. doi: 10.1097/SLA.0000000000000923. PMID 25203874
- [Background] Gulur P, Williams L, Chaudhary S, Koury K, Jaff M. Opioid tolerance--a predictor of increased length of stay and higher readmission rates. Pain Physician. 2014 Jul-Aug;17(4):E503-7. PMID 25054400
- [Background] Kessler ER, Shah M, Gruschkus SK, Raju A. Cost and quality implications of opioid-based postsurgical pain control using administrative claims data from a large health system: opioid-related adverse events and their impact on clinical and economic outcomes. Pharmacotherapy. 2013 Apr;33(4):383-91. doi: 10.1002/phar.1223. PMID 23553809
- [Background] Lembke A. Why doctors prescribe opioids to known opioid abusers. How cultural attitudes and financial disincentives affect the prescribing habits of physicians. Minn Med. 2013 Mar;96(3):36-7. No abstract available. PMID 23930467
- [Background] Volkow ND, Frieden TR, Hyde PS, Cha SS. Medication-assisted therapies--tackling the opioid-overdose epidemic. N Engl J Med. 2014 May 29;370(22):2063-6. doi: 10.1056/NEJMp1402780. Epub 2014 Apr 23. No abstract available. PMID 24758595
- [Background] Pugely AJ, Martin CT, Gao Y, Mendoza-Lattes S. Causes and risk factors for 30-day unplanned readmissions after lumbar spine surgery. Spine (Phila Pa 1976). 2014 Apr 20;39(9):761-8. doi: 10.1097/BRS.0000000000000270. PMID 24525993
- [Background] Hazratjee N, Agito M, Lopez R, Lashner B, Rizk MK. Hospital readmissions in patients with inflammatory bowel disease. Am J Gastroenterol. 2013 Jul;108(7):1024-32. doi: 10.1038/ajg.2012.343. PMID 23820989
- [Background] Centers for Disease Control and Prevention (CDC). CDC grand rounds: prescription drug overdoses - a U.S. epidemic. MMWR Morb Mortal Wkly Rep. 2012 Jan 13;61(1):10-3. PMID 22237030
- [Background] Bell JR. Australian trends in opioid prescribing for chronic non-cancer pain, 1986-1996. Med J Aust. 1997 Jul 7;167(1):26-9. doi: 10.5694/j.1326-5377.1997.tb138759.x. PMID 9236756
- [Background] Bot AG, Bekkers S, Arnstein PM, Smith RM, Ring D. Opioid use after fracture surgery correlates with pain intensity and satisfaction with pain relief. Clin Orthop Relat Res. 2014 Aug;472(8):2542-9. doi: 10.1007/s11999-014-3660-4. Epub 2014 Apr 29. PMID 24777731
- [Background] Herzig SJ, Rothberg MB, Cheung M, Ngo LH, Marcantonio ER. Opioid utilization and opioid-related adverse events in nonsurgical patients in US hospitals. J Hosp Med. 2014 Feb;9(2):73-81. doi: 10.1002/jhm.2102. Epub 2013 Nov 13. PMID 24227700
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Torrance N, Elliott AM, Lee AJ, Smith BH. Severe chronic pain is associated with increased 10 year mortality. A cohort record linkage study. Eur J Pain. 2010 Apr;14(4):380-6. doi: 10.1016/j.ejpain.2009.07.006. Epub 2009 Sep 1. PMID 19726210
- [Background] Pavon JM, Zhao Y, McConnell E, Hastings SN. Identifying risk of readmission in hospitalized elderly adults through inpatient medication exposure. J Am Geriatr Soc. 2014 Jun;62(6):1116-21. doi: 10.1111/jgs.12829. Epub 2014 May 6. PMID 24802165
- [Background] Muthuvel G, Tevis SE, Liepert AE, Agarwal SK, Kennedy GD. A composite index for predicting readmission following emergency general surgery. J Trauma Acute Care Surg. 2014 Jun;76(6):1467-72. doi: 10.1097/TA.0000000000000223. PMID 24854317
- [Background] Wilson GC, Cutler Quillin R 3rd, Sutton JM, Wima K, Shaw JJ, Hoehn RS, Paquette IM, Abbott DE, Shah SA. Factors related to readmission after major elective surgery. Dig Dis Sci. 2015 Jan;60(1):47-53. doi: 10.1007/s10620-014-3306-0. Epub 2014 Jul 27. PMID 25064214
- [Background] Anderegg SV, Wilkinson ST, Couldry RJ, Grauer DW, Howser E. Effects of a hospitalwide pharmacy practice model change on readmission and return to emergency department rates. Am J Health Syst Pharm. 2014 Sep 1;71(17):1469-79. doi: 10.2146/ajhp130686. PMID 25147171
- [Background] Tayne S, Merrill CA, Shah SN, Kim J, Mackey WC. Risk factors for 30-day readmissions and modifying postoperative care after gastric bypass surgery. J Am Coll Surg. 2014 Sep;219(3):489-95. doi: 10.1016/j.jamcollsurg.2014.03.054. Epub 2014 May 20. PMID 25151343